CLINICAL TRIAL: NCT00782912
Title: Is Postpartum Anemia an Independent Risk Factor for Development of Postpartum Depression?
Brief Title: Postpartum Anemia and Postpartum Depression
Acronym: PPADS
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 08-155
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Postpartum Depression
Keywords: postpartum anemia, postpartum depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Postpartum anemia (PPA) and Postpartum depression (PPD) are common afflictions affecting women after childbirth. Both disorders have a significant impact on women's health and functional status. Despite common symptoms and characteristics, a link between these entities has not been adequately studied. The objective of this study is to determine whether postpartum anemia is an independent risk factor for the development of postpartum depression. This prospective cohort study will include all women delivered by elective term cesarean delivery. Hemoglobin and iron levels will be measured, standardized questionnaires for assessment of PPD, functional status and lactation will be administered before discharge and at 3 & 6 weeks post partum. Hemoglobin levels at each time point will be analyzed for correlation with depressive symptoms, functional status and lactation success.

ELIGIBILITY:
Inclusion Criteria:

* Women after term elective cesarean section

Exclusion Criteria:

* age < 16 years, preterm (< 37 weeks) delivery, multiple gestation, symptomatic anemia necessitating blood transfusion, significant fetal anomalies or infant not discharged with mother for other reason, preexisting severe chronic maternal illness, preexisting maternal depression and/or current use of antidepressants, other psychiatric illness (e.g. bipolar disease, schizophrenia) or preexisting hemoglobinopathy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women after term elective cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2008-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Incidence of postpartum depression | 0-6 weeks postpartum

SECONDARY OUTCOMES:
Mean Edinburgh Postnatal Depression Scale results | 0-6 weeks postpartum
Functional status | 0-6 weeks postpartum
Lactation success | 0-6 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Howard Berger, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada